CLINICAL TRIAL: NCT05906368
Title: Hypotension Prediction Index to Predict Epidural-labor Analgesia Induced Hypotension -- Pilot Study
Brief Title: Hypotension Prediction Index to Predict Epidural-labor Analgesia Induced Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grace Lim, MD, MS (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor-Investigator, Grace Lim, MD, MS, Associate Professor, Chief Obstetric & Women's Anesthesiology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: STUDY23030009
Record Dates: First submitted 2023-05-08; First posted 2023-06-15 (Actual); Results first posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-08

CONDITIONS: Anesthesia, Epidural; Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Intervention Model Description: Participants are randomized to receive standard clinical care (SCC) blood pressure measurement or blood pressure monitoring of HPI via ClearSight with SCC.
Who Masked: Participant
Masking Description: Participants will wear both a conventional blood pressure cuff and the ClearSight finger cuff throughout the duration of the 4-hours post-epidural placement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Conventional Care (Sham Comparator): Patients are wearing both a conventional blood pressure cuff and the ClearSight finger cuff blood pressure monitoring system. Only measures from the conventional blood pressure cuff are sent/received by the clinical staff in the central and local nursing and anesthesia staff areas. The ClearSight monitoring system data is collected but not used by the clinical staff team for hypotensive monitoring.
  Interventions: Diagnostic Test: Standard of Care Blood Pressure Monitoring
- ClearSight Monitoring (Experimental): Patients are wearing both a conventional blood pressure cuff and the ClearSight finger cuff blood pressure monitoring system. Measures from BOTH the conventional blood pressure cuff and ClearSight monitoring system are sent/received by the clinical staff in the central and local nursing and anesthesia staff areas. ClearSight monitoring will add additional information regarding hypotensive events for clinical staff to respond to.
  Interventions: Diagnostic Test: ClearSight HPI Monitoring system; Diagnostic Test: Standard of Care Blood Pressure Monitoring

INTERVENTIONS:
Diagnostic Test: ClearSight HPI Monitoring system — Continuous blood pressure monitoring for precision hypotensive event response
  Arms: ClearSight Monitoring
Diagnostic Test: Standard of Care Blood Pressure Monitoring — Blood pressure (BP) monitoring using a conventional arm cuff and inflation after epidural anesthesia as standard procedure. Standard of care blood pressure monitoring includes measurement of blood pressure at the time of epidural test dose delivery, 3-minute cycles of BP monitoring for 30 minutes after epidural placement, and then BP monitoring every 15 minutes per existing clinical standards for at least 4-hours, or until delivery.

SUMMARY:
The purpose of this pilot trial is to examine the feasibility and ease of use of monitoring by ClearSight in laboring and delivering patients with the intent to compare time-to-treatment of hypotension between conventionally monitored patients (Group CM) and those receiving HPI (Group CM + HPI) monitoring by ClearSight, in a population of healthy laboring women who receive epidural analgesia.

DETAILED DESCRIPTION:
In a prospective study, we will achieve the following aims:

To determine the feasibility and ease of use of the ClearSight monitoring system in the labor-delivery room (LDR) in detecting and monitoring hypotensive events post-epidural labor analgesia placement.

To compare the Time-to-Treatment of hypotensive events between the conventionally monitored patients (Group CM) and those receiving HPI (Group CM + HPI) monitoring by ClearSight.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Age ≥ 18 years of age
* Planning vaginal delivery
* Receiving epidural labor analgesia (ELA)

Exclusion Criteria:

* Non-reassuring fetal tracing at the time of ELA request
* Contraindications to ELA
* Significant cardiac arrhythmias or aortic regurgitation
* Arrhythmia
* Treatment with antihypertensive medications
* Pre-eclampsia with or without severe features
* Preoperative infection
* Inability to use ClearSight device for any reason
* Non-English fluency
* Sustains unintentional dural puncture
* Incomplete data

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-04-18 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace Lim, MD, MSc, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Conventional Care | ClearSight Monitoring
Started | 17 | 17
Completed | 14 | 16
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Ineligibility criteria identified | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Care | ClearSight Monitoring | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (5.5) | 29.8 (5.7) | 29.6 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 12 | 13 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 32.4 (5.1) | 34.9 (6.3) | 33.7 (5.8)

OUTCOME MEASURES:

1. Primary Outcome: Time-to-treatment of Hypotension (Minutes)
Description: The difference in time between diagnosis of hypotension and treatment by clinical staff between CM and HPI groups
Time Frame: From epidural placement until 4-hours post-infusion start
Population: Only subjects with a hypotensive event were analyzed for this outcome measure (n=20)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Conventional Care | ClearSight Monitoring
Number analyzed (Participants) | 10 | 10
minutes | 21.8 (17.5) | 23.1 (17.6)

2. Primary Outcome: Ease of Use by Clinical Staff
Description: Clinical nurse reports of ease of use of ClearSight device. This outcome will be measured on a Likert Scale (0-4) with the options being: 0-Completely Disagree, 1-Disagree, 2-Neither agree nor disagree, 3-Agree, 4-Completely Agree. Outcome measure will be reported as count of participant's responses per category. For this scale, the objective was to obtain agreeable response feedback (score of 3 or 4). The specific question to measure ease of use by clinical staff was: "The ClearSight blood pressure monitoring device seems easy to use."
Time Frame: report at 4-hour post-infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Care | ClearSight Monitoring
Number analyzed (Participants) | 14 | 16
Participants
  Disagree | 1 | 1
  Neither agree nor disagree | 4 | 4
  Agree | 6 | 7
  Completely Agree | 3 | 4

3. Primary Outcome: Ease of Hypotension Detection by Clinical Staff
Description: Clinical nurse reports of ease of hypotension detection using ClearSight device. This outcome will be measured on a Likert Scale (0-4) with the options being: 0-Completely Disagree, 1-Disagree, 2-Neither agree nor disagree, 3-Agree, 4-Completely Agree. Outcome measure will be reported as count of participant's responses per category. For this scale, the objective was to obtain agreeable response feedback (score of 3 or 4). The specific question to measure ease of use by clinical staff was: "The ClearSight blood pressure monitoring device seems suitable."
Time Frame: report at 4-hour post-infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Care | ClearSight Monitoring
Number analyzed (Participants) | 14 | 16
Participants
  Disagree | 1 | 1
  Completely Agree | 4 | 3
  Neither agree nor disagree | 0 | 2
  Agree | 9 | 10

4. Primary Outcome: Satisfaction of ClearSight Use by Clinical Staff
Description: Clinical nurse reports of satisfaction of use of ClearSight device. This outcome will be measured on a Likert Scale (0-4) with the options being: 0-Completely Disagree, 1-Disagree, 2-Neither agree nor disagree, 3-Agree, 4-Completely Agree. Outcome measure will be reported as count of participant's responses per category. For this scale, the objective was to obtain agreeable response feedback (score of 3 or 4). The specific question to measure ease of use by clinical staff was: "The ClearSight blood pressure monitoring device meets my approval."
Time Frame: report at 4-hour post-infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Care | ClearSight Monitoring
Number analyzed (Participants) | 14 | 16
Participants
  Disagree | 1 | 0
  Completely Agree | 5 | 5
  Agree | 7 | 8
  Neither agree nor disagree | 1 | 3

5. Secondary Outcome: Total Time in Hypotension With Mean Arterial Pressure (MAP) <65 mmHg (in Minutes)
Description: Average number of minutes patients spent within hypotensive events for each group (CM and CM + HPI).
Time Frame: Epidural placement to 4-hours post-infusion start
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Conventional Care | ClearSight Monitoring
Number analyzed (Participants) | 14 | 16
minutes | 12.5 (19.3) | 7.7 (9.5)

6. Secondary Outcome: Nausea (Yes/No)
Description: Proportion of patients by group reporting nausea within 4-hours of post-epidural placement
Time Frame: Epidural placement to 4-hours post-infusion start
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Care | ClearSight Monitoring
Number analyzed (Participants) | 14 | 15
Participants
  Yes Nausea | 5 | 7
  No Nausea | 9 | 8

7. Secondary Outcome: Vomiting (Yes/No)
Description: Proportion of patients by group reporting Vomiting within 4-hours of post-epidural placement
Time Frame: Epidural placement to 4-hours post-infusion start
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Care | ClearSight Monitoring
Number analyzed (Participants) | 14 | 16
Participants
  Yes Vomiting | 3 | 0
  No Vomiting | 11 | 16

8. Secondary Outcome: Total Phenylephrine, mg
Description: Average phenylephrine dose(s) given to patients in CM and CM+HPI groups
Time Frame: Epidural placement to 4-hours post-infusion start
Population: Only subjects with a hypotensive event and received phenylephrine were analyzed for this outcome measure (n=9)
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Conventional Care | ClearSight Monitoring
Number analyzed (Participants) | 6 | 3
mg | 223.3 (242.1) | 506.7 (410.5)

9. Secondary Outcome: Total Ephedrine, mg
Description: Average ephedrine dose(s) given to patients in CM and CM+HPI groups
Time Frame: Epidural placement to 4-hours post-infusion start
Population: Only subjects with a hypotensive event and received epinephrine were analyzed for this outcome measure (n=19)
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Conventional Care | ClearSight Monitoring
Number analyzed (Participants) | 10 | 9
mg | 29.8 (26.4) | 23.3 (23.6)

10. Secondary Outcome: Total Intravenous Fluids, mL
Description: Average volume of fluids given to patients in CM and CM+HPI groups
Time Frame: Epidural placement to 4-hours post-infusion start
Population: Only subjects with a hypotensive event and received IV fluids were analyzed for this outcome measure (n=16)
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Conventional Care | ClearSight Monitoring
Number analyzed (Participants) | 9 | 7
mL | 550.0 (169.6) | 535.7 (94.5)

11. Secondary Outcome: Total Number of Reported Changes in Fetal Heart Rate Category (From Healthy to Deceleration or Excelleration)
Description: Total number of participants who experienced changes in fetal heart rate category (any)
Time Frame: Epidural placement to 4-hours post-infusion start
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Care | ClearSight Monitoring
Number analyzed (Participants) | 14 | 15
Participants
  Yes - Changes in fetal heart rate | 8 | 6
  No - Changes in fetal heart rate | 6 | 9

12. Secondary Outcome: Fetal Heart Rate Decelerations Within 1 Hour of Initiation of ELA
Description: Percentage of patients who experience any fetal heart rate deceleration event [Presence (Yes) or absence (No)] within 1-hour of epidural placement.
Time Frame: Epidural placement to 1-hour post-infusion start
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Care | ClearSight Monitoring
Number analyzed (Participants) | 14 | 15
Participants
  Yes | 5 | 5
  No | 9 | 10

ADVERSE EVENTS:
Time Frame: 36+ weeks gestation to 12-weeks postpartum per subject
Arm/Group | Conventional Care | ClearSight Monitoring
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 0/14 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-07): https://cdn.clinicaltrials.gov/large-docs/68/NCT05906368/Prot_SAP_002.pdf
  • Informed Consent Form (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/68/NCT05906368/ICF_001.pdf